CLINICAL TRIAL: NCT01963117
Title: Effectiveness of the Combined Whole Liver Irradiation (WLI) and Hyperthermia for Unresectable Chemoresistant Multiple Liver Metastasis From Gastrointestinal Tract Cancer: Prospective Phase II Trial
Brief Title: Effectiveness of the Combined WLI and Hyperthermia for GI Cancer Liver Metastasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2013-06-040
Record Dates: First submitted 2013-09-25; First posted 2013-10-16 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2014-08

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined hypertermia and RT (Experimental): Combined hypertermia and radiothearpy
  Interventions: Radiation: Combined hyperthermia and radiation therapy

INTERVENTIONS:
Radiation: Combined hyperthermia and radiation therapy

SUMMARY:
The standard treatment of unresectable liver metastasis in gastrointestinal tract cancer is chemotherapy, but considerable portion of the patients progressed and most of the liver is converted to metastatic tumor lesions. Significant quality of life decrement was detected in those patients, especially in patients suffered severe symptoms Several studies reported that whole liver RT (WLRT) can be used effectively to control severe symptoms from unresectable liver metastasis in gastrointestinal tract cancer patients. However, it is well known fact that the liver is a very sensitive to RT. Despite symptom palliation is obtained after 20 to 30 Gy RT but only in small subset of patients get local control. In this aspect, the combined with radiosensitizer with WLRT is considered to enhance RT effect to palliate symptom and control local tumor progression, and increase the quality of life ultimately.

It is reported that hyperthermia is considered as the most valuable radiosensitizer in cancer treatment, theoretically. Based on those studies, we start this prospective study to investigate the effect of combination treatment of WLRT and hyperthermia on quality of life in the patients with unresectable chemoresistant liver metastasis from gastrointestinal tract cancer.

DETAILED DESCRIPTION:
1.1 gastrointestinal tract cancer liver metastasis Most mortality of the gastrointestinal tract cancer patients is related with distant metastasis, especially liver is the main site. It has been estimated that 25% of colorectal cancer patients have hepatic metastases at diagnosis, and another 50% will have their tumor recurrence in the liver within 5 years.

Selected patients who had oligo (usually 2 to 3) or isolated liver metastases resected curatively and have yielded 5-year survival rates of 50% to 60%, showing that local therapy has the potential to cure. It is only possible in less than 25% of all patients with hepatic metastasis because of medical and/or surgical reasons, furthermore two-thirds of resected patients showed ultimately liver recurrence within 2 years.

The standard treatment of unresectable liver metastasis in gastrointestinal tract cancer is chemotherapy, but considerable portion of the patients progressed and most of the liver is converted to metastatic tumor lesions. Significant quality of life decrement was detected in those patients, especially in patients suffered severe symptoms

1.2 Radiation therapy (RT) for liver metastasis Several studies reported that whole liver RT (WLRT) can be used effectively to control severe symptoms from unresectable liver metastasis in colorectal cancer patients. However, it is well known fact that the liver is a very sensitive to RT. The radiation induced liver disease (RILD), dreadful complication without special treatment method and subset of patients could be dead, can be developed as low as 30 gray (Gy). Despite symptom palliation is obtained after 20 to 30 Gy RT but only in small subset of patients get local control. In this aspect, the combined with radiosensitizer with WLRT is considered to enhance RT effect to palliate symptom and control local tumor progression, and increase the quality of life ultimately.

1.3 Hyperthermia It is reported that hyperthermia is effective in S phase, Low oxygen partial pressure (pO2), low hydrogen ion concentration (pH), and low perfusion site which are known as radio-resistant. Because of these characteristics, it considered as the most valuable radiosensitizer in cancer treatment, theoretically. Furthermore, mild hyperthermia (41 to 41.5 ºC) can promote tumor reoxygenation.

1.4 Purpose of this study Based on those studies, we start this prospective study to investigate the effect of combination treatment of WLRT and hyperthermia on quality of life in the patients with unresectable chemoresistant liver metastasis from gastrointestinal tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1 Patients must have a diagnosis of pathologic proven gastrointestinal tract cancer
* 2 Unresectable and unsuitable to other local modalities
* 3 Not responded and/or unsuitable to chemotherapy
* 4 Eastern Cooperative Oncology Group ECOG) performance status 0 to 3
* 5 Assessment by colorectal tumor board (surgeon, radiation oncologist and medical oncologist participated)
* 6 Age ≥ 20
* 7 Agreement of study-specific informed consent
* 8 Blood work requirements

  * Absolute neutrophil count (ANC) ≥ 1,500 /mm3, Platelet ≥ 50,000/mm3, Hgb ≥ 8 g/dl
  * Liver function test(LFT): Total bilirubin<3.0 mg/dL, International normalized ratio(INR) < 1.7, Albumin ≥ 2.8g/dL, Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT)< 6 X normal
  * Serum creatinine < 1.5 X normal, or Creatinine clearance rate (CCr) ≥ 60 mL/min
* 9 Child-Pugh score 10 or less within 1 week before WLI
* 10 Childbearing potential woman, consent contraception at least 6 months
* 11 Stable breathing more than 5 minutes

Exclusion Criteria:

* 1 Life expectancy less than 8 weeks
* 2 Pregnant and/or breastfeeding woman
* 3 Previous upper abdominal RT history
* 4 Uncontrolled ascites or hepatic encephalopathy
* 5 Unstable respiration due to pleural effusion, chronic obstructive pulmonary disease COPD) etc

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hee Chul Park, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Hypertermia and RT: Combined hyperthermia and radiation therapy
Period: Overall Study
Arm/Group | Combined Hypertermia and RT
Started | 11
Completed | 10
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: HCC patients who will receive combination treatment with transarterial chemoembolization, radiotherapy, and hyperthermia
Groups:
- CERT: Combination treatment with transarterial chemoembolization, radiotherapy, and hyperthermia
Arm/Group | CERT
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 56 [35 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  South Korea | 11
Child Pugh Class [Number; unit: participants] — Child Pugh Class A; score 5 to 6 Child Pugh Class B; score 7 to 10 Child Pugh Class Cl score 11 to 18
  Total range of score is 5 to 18 with higher scores/increased scores indicate greater severity of poor liver function.
  participants
    Child Pugh Class A | 9
    Child Pugh Class B | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Local Tumor Progression After Combined Hyperthermia and RT
Description: Local progression will be defined as more than 20% size increase of metastatic lesions or new metastatic lesion in liver. Time to local tumor progression will be measured from the date of RT start to the date of local progression or last follow-up visit.
Time Frame: Patient will be evaluated after combined hyperthermia and RT until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 19 months.
Population: Patients who underwent combined hyperthermia and radiation therapy
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Combined Hypertermia and RT
Number analyzed (Participants) | 10
Months | 18.5 [15.1 to 21.9]

2. Secondary Outcome: Objective Response Rate of Combined Hyperthermia and RT
Time Frame: Response will be evaluated at 3 month after combined hyperthermia and RT. Modified RECIST will be used to define resopnse.
Measure: Number; unit: participants
Arm/Group | Combined Hypertermia and RT
Number analyzed (Participants) | 10
participants | 10

3. Secondary Outcome: Change in the Grade of Quality of Life at 3 Months From That Before the Combined Hyperthermia and RT
Description: To measure the quality of life, European Organisation for Research and Treatment of Cancer (EORTC)- quality of life questionnaire (QLQ) 30 and Functional Assessment of Cancer Therapy-Hepatobiliary will be used. (grade 1 to 4, 1; not at all, 2; a little, 3; quite a bit, 4; very much)
Time Frame: Quality of life will be ssessed at baseline and 3 months after combined hyperthemica and RT, data reported 3 months after combined hyperthemica and RT with grade from 1 to 4.
Population: European Organisation for Research and Treatment of Cancer (EORTC)- quality of life questionnaire (QLQ) 30 and Functional Assessment of Cancer Therapy-Hepatobiliary will be used from grade 1 to 4.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Combined Hypertermia and RT
Number analyzed (Participants) | 4
score on a scale | -2 [-3 to 3]

4. Secondary Outcome: Local Tumor Progression Free Survival Rate After Combined Hyperthermia and RT
Description: Local progression will be defined as more than 20% size increase of metastatic lesions or new metastatic lesion in liver. Local progression free survival will be measured from the date of RT start to the date of local progression or last follow-up visit.
Time Frame: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Combined Hypertermia and RT
Number analyzed (Participants) | 10
Months | 18.5 [15.1 to 21.9]

5. Secondary Outcome: Adverse Event After Combined Hyperthermia and RT.
Description: All grade III or higher toxicities (repeated measure)
Time Frame: Adverse event will be evaluated at 3 month. The common terminology criteria for adverse events (CTCAE) version 4.0 will be used.
Measure: Number; unit: participants
Arm/Group | Combined Hypertermia and RT
Number analyzed (Participants) | 10
participants | 1

6. Secondary Outcome: Overall Survival Rate After Combined Hyperthermia and RT
Description: Overall survival will be measured from the date of RT start to the date of death or last follow-up visit.
Time Frame: Pathient will be evaluated at 3 month after combined hyperthermia and RT.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Combined Hypertermia and RT
Number analyzed (Participants) | 10
Months | 18 [15.1 to 19]

ADVERSE EVENTS:
Arm/Group | Combined Hypertermia and RT
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Hypertermia and RT (N=11)
Death (Respiratory, thoracic and mediastinal disorders) | 4 (5) — Pneumonitis outside RT field

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes